CLINICAL TRIAL: NCT03608579
Title: ASCLEPIOS Autologous Stem CelL Expansion and Prospective Injection for Osteoarthritic Hip Symptoms
Brief Title: Autologous Culture Expanded Adipose Derived MSCs for Treatment of Painful Hip OA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron Krych, Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-000015
Record Dates: First submitted 2018-07-10; First posted 2018-08-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Injection (Experimental): Single administration of Autologous Adipose Derived Mesenchymal Stromal Cells into the hip by single ultrasound guided injection
  Interventions: Drug: Autologous Adipose Derived Mesenchymal Stromal Cells
- Two Injections (Experimental): Two-dose administration (2 x ultrasound guided injections) of Autologous Adipose Derived Mesenchymal Stromal Cells into the hip with one month interval between doses
  Interventions: Drug: Autologous Adipose Derived Mesenchymal Stromal Cells

INTERVENTIONS:
Drug: Autologous Adipose Derived Mesenchymal Stromal Cells — Human, autologous, culture expanded, adipose derived, mesenchymal stromal cells (AMSCs) produced on site in the Mayo Clinic Human Cellular Therapy Laboratory using current good manufacturing practices
  Other Names: ASCLEPIOS

SUMMARY:
Will injection(s) of autologous culture-expanded AMSCs be safe and efficacious for treatment of painful Hip OA, and if so, which dosing regimen is most effective?

DETAILED DESCRIPTION:
This phase I study will enroll 24 subjects with mild to moderate osteoarthritis of the hip. Subjects will receive either a single dose of 30 million autologous culture-expanded adipose-derived mesenchymal stromal cells (AMSCs), or two doses of AMSCs (with one month interval between doses) via ultrasound guided intra-articular hip injection. Patients will be followed for 24 months past their last injection to determine the local and systemic safety of single and two-dose injections of AMSCs in the treatment of symptomatic hip OA.

ELIGIBILITY:
Inclusion Criteria

To be eligible for inclusion into this study, the subjects must fulfill all of the following criteria:

1. Male or female ages 18-65 years

   • Persons of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 1 year following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit
2. Persons becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded.
3. Chronic (> 3 months), unilaterally symptomatic, primary hip OA. Patients with episodes of contralateral hip pain that is asymptomatic at the time of enrollment will be eligible for inclusion. However, as outlined in the primary study endpoints, patients with previous episodes of contralateral hip pain who experience a repeat episode of contralateral pain similar to their established pattern of pain during the course of the trial will not be considered as having experienced an adverse event.
4. Radiographic hip OA of Tönnis Grade 1 - 2, accompanied by at least mild sclerosis and joint space narrowing, as agreed upon by two study co-investigators without underlying structural hip abnormalities
5. Previous 6 week or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications or injection therapy (e.g. cortisone)
6. Able to routinely walk without assistance (e.g. cane, walker)
7. Clinically stable target hip
8. No surgery planned in the target hip for at least 12 months following the last injection
9. Completed general physical and well-being evaluation with primary care provider within 12 months of enrollment
10. Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including fat harvesting, laboratory tests, diagnostic imaging, and follow-up visits and assessments
11. Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure

Exclusion Criteria

To be eligible for inclusion in this study, the subjects must not meet any of the following criteria:

1. Pregnant or nursing, or planning on becoming pregnant during the study period
2. Congenital or acquired malformation of the target hip resulting in significant deformity or leading to problems with the study treatment or analysis of the results
3. Significant structural deformity, including large cam lesion (alpha angle greater than 55 degrees) or moderate dysplasia (defined as lateral center edge angle less than 18 degrees).
4. Injections of any kind into the target hip within 3 months prior to study enrollment
5. Locking, catching, give-away or another major mechanical symptoms of the target hip
6. History of intra-articular infection in the target hip
7. History of superficial infection in the target hip within 6 months of study enrollment, or evidence of current superficial infection affecting the target hip
8. History of falls requiring medical attention, or gait instability
9. Clinically significant abnormal hematology (complete blood count with differential), blood chemistry, or urinalysis screening laboratory results.
10. Body mass index (BMI) > 35 kg/m2
11. Taking anticoagulant medications (e.g. warfarin, heparin or clopidogrel) which may pose a clinically-significant contraindication to intra-articular injection.
12. Taking herbal therapies or supplements within 4 weeks of enrollment or unwilling to avoid use of herbal therapies or supplements until at least 30 days following completion of the study drug treatment cycle (includes, but not limited to chondroitin sulfate, diacerein, n-glucosamine and capsaicin)
13. Taking non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) without a stable dosing regimen for at least 4 weeks before baseline evaluation, or anticipating not remaining on a stable dose until at least 30 days following completion of the study drug treatment cycle
14. Use of electrotherapy or acupuncture for OA, unless there is a stable regimen for at least 4 weeks before baseline assessment
15. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment
16. On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
17. Current tobacco product use, including nicotine patch or other nicotine products
18. Clinically significant systemic inflammatory, rheumatological or connective tissue disorder including but not limited to rheumatoid arthritis, systemic sclerosis, system lupus erythematosus, and Ehlers-Danlos Syndrome
19. Clinically significant rheumatological or inflammatory disease of the hip or chondrocalcinosis/calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the hip associated with juxta-articular Paget's disease of the femur or pelvis, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's hip joint, villonodular synovitis, and synovial chondromatosis
20. Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis
21. Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurologic (e.g. stroke, TIA) renal, hepatic, orthopedic (e.g. surgery on other weight bearing joints that will interfere with study, osteoporosis, acute lower body fractures), or endocrine disease (e.g. diabetes).
22. Vascular or neurological disorder affecting the either lower limb which poses clinical significance to the safe delivery of intra-articular therapy.
23. History of cancer/malignancy with the exception of adequately treated basal cell or squamous cell carcinoma of the skin not associated with the target hip
24. History of clinically significant blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy
25. Participation in a study of an experimental drug or medical device within 3 months of study enrollment
26. Known allergy to local anesthetics of other components of the study drug
27. Any contraindication to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures
28. History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 30 days of study entry
29. Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Nature, incidence and severity of adverse events (AEs) | For a period of 2 years following last injection
  Defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship.
  Methods i. Spontaneous subject reports ii. Subject interview by study personnel iii. Clinical examination during face-to-face clinic follow-ups

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) for pain in the target hip following completion of treatment cycles | Baseline, 6 weeks, 6 months, 12 months post-treatment cycle
  100 mm Visual Analog Scale. Range: 0 to 100 mm. Lower is better, higher is worse.
Change in Tegner activity scale in the target hip following completion of treatment cycles | Baseline, 6 weeks, 6 months, 12 months post-treatment cycle
  Tegner activity scale (Level 0 to Level 10). Higher is better, lower is worse.
Change in modified Harris Hip Score (mHHS) in the target hip following completion of treatment cycles | Baseline, 6 weeks, 6 months, 12 months post-treatment cycle
  modified Harris Hip Score (mHHS). Score 0 to 100. Higher is better, lower is worse.
Change in Hip disability and osteoarthritis Outcome Score (HOS) in the target hip following completion of treatment cycles | Baseline, 6 weeks, 6 months, 12 months post-treatment cycle
  Hip disability and osteoarthritis Outcome Score (HOS). Score 0 to 100. Higher is better, lower is worse.
Change in radiographic joint morphology | Baseline, 6 months, and 12 months post-treatment cycle
  Evaluation of joint morphology on hip X-rays, including standing antero-posterior, lateral, and false profile
Change in cartilage thickness | Baseline, 6 months, and 12 months post-treatment cycle
  Cartilage thickness on MRI
Change in cartilage volume | Baseline, 6 months, and 12 months post-treatment cycle
  Cartilage volume on MRI
Change in cartilage morphology | Baseline, 6 months, and 12 months post-treatment cycle
  Cartilage morphology on MRI
Change in subchondral bone morphology | Baseline, 6 months, and 12 months post-treatment cycle
  Subchondral bone morphology (i.e. edema) on MRI
Change periarticular soft-tissues | Baseline, 6 months, and 12 months post-treatment cycle
  Evaluate periarticular tissues on MRI (i.e. visible synovitis)
Change in synovial fluid biomarkers within the target hip | Baseline at the time of AMSC injection, At time of second injection (1 month status post first injection) in 2-injection group
  Synovial fluid from attempted aspiration at the time of injection (and re-injection for the two injection cohort) will be analyzed for cells, cytokines, growth factors, and other similar biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Krych, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials